CLINICAL TRIAL: NCT00719992
Title: Diagnostic Value of HS-CRP in Stable Angina Patients With Positive Exercise Test as Compared With Coronary Angiography.
Brief Title: Diagnostic Value of HS-CRP in Stable Angina.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Dr Javad Kojuri, Shiraz University of medical sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 4543
Record Dates: First submitted 2008-07-18; First posted 2008-07-22 (Estimated); Last update posted 2008-07-22 (Estimated); Status verified 2008-07

CONDITIONS: Stable Angina; Positive ETT
Keywords: Exercise tolerance test; HS-CRP; Coronary angiography; Patients
MeSH Terms: conditions — Angina, Stable

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): positive ETT, High HS-CRP
  Interventions: Procedure: coronary angiography
- 2 (Active Comparator): positive ETT, Low HS-CRP
  Interventions: Procedure: coronary angiography

INTERVENTIONS:
Procedure: coronary angiography — effect of level of HS-CRP

SUMMARY:
The aim of this study was to assess the amount of additive value of HS-CRP levels to a positive exercise tolerance test (ETT) in predicting coronary artery disease (CAD) using coronary angiography as the gold standard. The investigators concluded that HS-CRP can be used as a single predictor of coronary vessel involvement in patients with stable angina and positive ETT.

DETAILED DESCRIPTION:
the investigators included 97 patients with positive ETT and stable angina and saw that Hs-CRP is the only predictor of severity of CAD as compared with coronary angiography in stable angina patients.

ELIGIBILITY:
Inclusion Criteria:

* Stable angina
* Positive ETT

Exclusion Criteria:

* Unability to perform ETT
* Contraindications for ETT and angiography study

Ages: 43 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2006-04; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
significant coronary lesion

SECONDARY OUTCOMES:
severity of CAD

CONTACTS AND LOCATIONS:
Overall Officials: javad kojuri, M.D., Study Director — Shiraz University of Medical Sciences
Locations (1):
- Cardiology Ward Shiraz University of Medical Sciences, Shiraz, Fars, Iran